CLINICAL TRIAL: NCT00811343
Title: Impact of New Immunological Diagnosis Tests of Latent Tuberculosis in Adults Patients Who Need Anti TNF Therapy.
Brief Title: Impact of New Immunological Diagnosis Tests of Latent Tuberculosis Before Anti TNF Therapy
Acronym: ETAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P070310; 2008-A00744-51 (Other: IDRCB)
Record Dates: First submitted 2008-12-18; First posted 2008-12-19 (Estimated); Last update posted 2014-01-07 (Estimated); Status verified 2014-01

CONDITIONS: Tuberculosis
Keywords: anti TNF Therapy; Tuberculosis; Tuberculin test; QFTB-G; T-SPOT.TB; Need anti TNF Therapy
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Biological: QFTB-G and T-SPOT.TB tests

INTERVENTIONS:
Biological: QFTB-G and T-SPOT.TB tests — QFTB-G and T-SPOT.TB test before TST
  Other Names: There are no arms currently listed for this study.

SUMMARY:
Tuberculosis is a current infection during anti TNF therapy. After infectious contact, some patients will develop tuberculosis and some will only be infected without symptoms, they have Latent Tuberculosis Infection (LTBI) wich can reactivate later. In order to prevent this tuberculosis reactivation, LTBI diagnosis screening is preconised in patients who need anti TNF therapy. This diagnosis is made till now by the tuberculin skin test (TST) but this test is not specific of TB. New blood tests (QFTB-G and T-SPOT.TB) specific to MTB infection are now available.

The primary endpoint of this study is the evaluation of the theoric therapeutic impact of the use of new tests for diagnosis of LTBI in patients before anti TBF therapy

DETAILED DESCRIPTION:
Detailed description :

Principal outcome: Therapeutic impact of the use of new tests for diagnosis of LTBI in patients before anti TBF therapy

Secondary outcomes :

* medico-economic impact of replacement of TST by QFTB-G and T-SPOT.TB tests in LTBI screening in patients before anti TNF therapy.
* concordance of QFTB-G and T-SPOT.TB tests results with TST
* Concordance between QFTB-G and T-SPOT.TB tests and evaluation of indetermined tests.
* concordance of QFTB-G and T-SPOT.TB tests results with patient disease.
* concordance of QFTB-G and T-SPOT.TB tests results with TST in patients with LTBI determinated by clinical or radiological observation
* Impact of geographical, disease and treatment in patients with LTBI determinated by clinical or radiological observation
* Identify the original characteristic and maximal impact therapeutic of QFTB-G and T-SPOT.TB test

Analysed criteria :

* therapeutic impact
* Patients percentage with different therapeutic outcome based on usual recommendations medico-economic
* Medico-economic impact :impact of both tests as early and late cost - efficacy

Statistic :

* Primary criteria : Percentage of patients for whom therapeutic would have been changed by QFTB-G and T-SPOT.TB tests results compared to usual diagnosis strategy.
* Secondary criteria : Concordance of QFTB-G and T-SPOT.TB tests with TST Concordance between both QFTB-G and T-SPOT.TB tests .

  400 patients Timing : inclusions : 1 years

ELIGIBILITY:
Inclusion Criteria:

* 18 years old
* Patient with rheumatoid arthritis or Ankylosing spondylitis or Crohn's disease
* Patient without Anti TNF treatment and who need one by infliximab, adalimumab or etanercept
* Consent signed
* Patient with social right
* Patient who have been examined

Exclusion Criteria:

* Pregnancy and breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 430 (Actual)
Dates: Start 2008-12; Primary Completion 2010-12 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Therapeutic impact | 12 months

SECONDARY OUTCOMES:
medico-economic impact | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Mariette, Pr, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Bicêtre hospital, Le Kremlin-Bicêtre, France

REFERENCES:
- [Derived] Freund R, Granger B, Francois C, Carcelain G, Ravaud P, Mariette X, Fautrel B. Cost-effectiveness analysis of strategies using new immunological diagnostic tests of latent tuberculosis infection before TNF-blockers therapy. Presse Med. 2018 Feb;47(2):e9-e13. doi: 10.1016/j.lpm.2017.09.029. Epub 2018 Feb 23. PMID 29478790
- [Derived] Mariette X, Baron G, Tubach F, Liote F, Combe B, Miceli-Richard C, Flipo RM, Goupille P, Allez M, Salmon D, Emilie D, Carcelain G, Ravaud P. Influence of replacing tuberculin skin test with ex vivo interferon gamma release assays on decision to administer prophylactic antituberculosis antibiotics before anti-TNF therapy. Ann Rheum Dis. 2012 Nov;71(11):1783-90. doi: 10.1136/annrheumdis-2011-200408. Epub 2012 Jan 17. PMID 22258485